CLINICAL TRIAL: NCT06062030
Title: Efficacy and Safety of DWJ1609 for Bowel Cleansing Before Colonoscopy; a Prospective, Randomized, Single-blinded (Investigator), Parallel, Multi-center, Active-control, Non-inferiority, Phase 3 Clinical Trial
Brief Title: Efficacy and Safety of DWJ1609 for Bowel Cleansing Before Colonoscopy;
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DWJ1609301
Record Dates: First submitted 2023-08-29; First posted 2023-10-02 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Colonoscopy
Keywords: HCS; Bowel Cleansing

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Single-blinded (Investigator),
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test group (Experimental): Investigational Products (DWJ1609) Number of tablets: 20 tablets in total Drinking water: 2,550 mL in total
  The day before the colonoscopy [Day 1] ▶ Common: Eat a light breakfast the day before the examination, or take only clear fluids.
  Take 10 tablets of DWJ1609 with 425 mL of water in the early evening (18:00-20:00) the day before the test, followed by 2 more doses of 425 mL of water for 1 hour (takes a total of 1,275 mL of water).
  On the day of colonoscopy [Day 2]
  ▶ Common: On the day of the examination, only clear liquids should be taken before the examination. Complete the clinical trial medication and additional water intake at least 2 hours prior to the test or at the time indicated by the tester In the evening before the test, take 10 additional DWJ1609 tablets with 425 mL of water in the morning (04:00~08:00), 10 to 12 hours after taking DWJ1609, followed by 2 more doses of 425 mL of water for 1 hour (Total 1,275 mL of water).
  Interventions: Drug: DWJ1609
- control group (Active Comparator): Control Products (DWC202304) Number of tablets: 28 tablets in total Drinking water: 2,550 mL in total
  The day before the colonoscopy [Day 1] Take 14 tablets of DWC202304 with 425 mL of water in the early evening (18:00 to 20:00) the day before the test, followed by 2 more doses of 425 mL of water for 1 hour (takes a total of 1,275 mL of water).
  On the day of colonoscopy [Day 2]
  ▶ Common: On the day of the examination, only clear liquids should be taken before the examination. Complete the clinical trial medication and additional water intake at least 2 hours prior to the test or at the time indicated by the tester In the evening before the test, take 14 additional DWC202304 tablets with 425 mL of water in the morning of the test (04:00~08:00), 10 to 12 hours after taking DWC202304, and then take 425 mL of water twice for 1 hour (total 1,275 mL of water).
  Interventions: Drug: DWC202304

INTERVENTIONS:
Drug: DWJ1609 — Drug of test group
  Arms: test group
Drug: DWC202304 — Drug of control group
  Other Names: Orafang Tab
  Arms: control group

SUMMARY:
Phase of Development : III

Sponsor : DAEWOONG PHARMACEUTICAL

Study Sites and Principal Investigator : Dong ll Park M.D. Ph.D , Gastroenterology Kangbuk Samsung Hospital and other 6 study sites

Study Period : From the protocol approval date (institutional review board, IRB) 24 Months

Investigational product :

Investigational Products DWJ1609 (sodium sulfate potassium sulfate, Magnesium Sulfate Anhydrous , simethicone, sodium picosulphate)

Control Products DWC202304 (sodium sulfate potassium sulfate, Magnesium Sulfate Anhydrous , simethicone)

Target Diseases : A person who needs treatment before colonoscopy (X-ray, endoscopy)

Number of Subjects : 214 Subjects in total (85 subjects per group, 2 groups in total, considering a 20% dropout rate)

DETAILED DESCRIPTION:
Study Methodology :

Test subjects evaluated as suitable for participation in clinical trials are randomly assigned at a 1:1 ratio to the test group (DWJ1609) and the control group (DWC202304), and clinical trial drugs are distributed for each administration group.

Subjects take the distributed clinical trial drugs as split-dose in the early evening of the day before colonoscopy (Day 1) and in the morning of the day of examination (Day 2) Test subjects visit the clinical trial institution after completing all clinical trial drugs at least 2 hours before colonoscopy (Visit 2).

All test subjects undergo colonoscopy in the morning, and the tester takes an image of all colonoscopy processes according to a separate manual.

For safety evaluation, subjects will conduct a phone visit 2 days after colonoscopy (±1 day) (Visit 3) and a regular visit 7 days after (±1 day) (Visit 4). If additional confirmation is required in the electrocardiogram or laboratory test results at the discretion of the tester, a follow-up visit can be conducted after 28 days (±2 days) (Visit 5).

I

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women 19 years of age or older as of the date of consent in writing
2. a prospective colonoscopy patient
3. 19 kg/㎡ ≤ BMI < 30 kg/㎡
4. A person who voluntarily agrees to participate in this clinical trial and signs a written agreement Abbreviation: BMI = body mass index

Exclusion Criteria:

1. A person who undergoes colonoscopy for the following therapeutic purposes (1) balloon dilatation of the stenosis area (2) non-toxic giant colon or decompression of the S-phase colitis (sigmoid volvulus) (3) Removal of foreign substances (4) Vascular dysplasia, ulcer, tumor and treatment of bleeding after polypectomy (5) Treatment for stenosis or tumor bleeding (palliative treatment)
2. A person whose past history has been confirmed during a screening visit (1) Severe heart disease (insecurity angina, acute myocardial infarction, acute heart failure, cardiomyopathy, etc.) or acute respiratory failure within 24 weeks prior to screening (2) Epilepsy or seizures within 96 weeks prior to screening (3) Clinically significant intestinal surgical history regardless of duration (e.g., colon premature surgery, colon resection, etc.)

   a. However, appendectomy and hemorrhoids are excluded
3. A person who has been identified or suspected of the following comorbidities during a screening visit (1) active intestinal hemorrhage (2) gastrointestinal obstruction (intestinal obstruction, gastrointestinal obstruction, etc.), gastrointestinal perforation, gastric discharge disorder (gastrointestinal paralysis, gastric congestion, etc.) (3) Inflammatory bowel disease (ulcerative colitis, Crohn's disease, toxic colitis, toxic colitis, etc.) (4) Gastrointestinal ulcers, colorectal mucosal ulcers, ischemic colitis (5) an acute abdominal condition requiring surgery (6) A person who has been identified with the following major cardiovascular diseases

   ① congestive heart failure

   ② NYHA functional classification III or IV

   ③ Clinically significant arrhythmia identified by ECG, QTcFb delay (Male > 450 msec, Female > 470 msec) etc.

   b. QTc interval corrected by Fridericia's formula (7) Despite adequate medication, uncontrolled hypertension (SBP > 170 mmHg and DBP > 100 mmHg) (8) Diabetes undergoing insulin treatment or in need of insulin treatment (9) Clinically significant electrolyte abnormalities (sodium, potassium, calcium, magnesium, chloride, bicarbonate, phosphate etc.) (10) Those who are at risk of dehydration (transverse fusion, ascites, etc.) (11) Severe renal impairment (eGFRc < 30 mL/min/1.73m2) c. MDRD-eGFR (mL/min/1.73m2) = 186 × (serum creatinine concentration)-1.154 × (age)-0.203 (× 0.742, Female) (12) Child-Pugh class B or C (13) ALT or AST > three times the normal upper limit of the trachea (14) Severe nausea or vomiting that makes it difficult to participate in clinical trials (15) Active infection or high fever above 38℃ (except acute upper respiratory tract infection or local skin infection) (16) Active hepatitis B or C d. Defined as HBsAg positive during screening e. Defined as HCV Ab positive during screening (17) Test results of HIV antibodies and antibody test results
4. A person who is administering the following drugs during a screening visit or is expected to be administered by the time of completion of a colonoscopy (Day 2; Visit 2) (1) Constipation patients who are regularly administered laxatives or gastrointestinal motility promoters within 12 weeks prior to screening (e.g., two to three times a week or more) (2) Administration of laxatives, enema, simethicone, 5HT4 receptor agonist, iron preparation, opioid excluding clinical trial drugs within 7 days of clinical trial drug administration (Day 1)
5. A person who is hypersensitive to the ingredients of a clinical trial drug
6. a pregnant woman or a lactating woman
7. Fertility women and men who have a pregnancy plan or do not agree to perform appropriate contraception during the clinical trial. Appropriate contraception in this trial is as follows

   * hormonal contraceptive
   * implantation of intrauterine device or intrauterine system
   * Infertility procedures/surgery (e.g., bilateral ovarian ligation, vasectomy)
8. A person who has participated in another clinical trial/medical device clinical trial within 4 weeks of screening and has received/treated clinical trial medication/medical device
9. For other reasons, the tester determines that he/she is unfit to be tested for this clinical trial (e.g., clinically significant blood coagulation disorder, mental illness, dementia, drug or alcohol abuse history, oral administration of clinical trial drugs)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
The successful cleaning rate of the Harefield Cleansing Scale (HCS) phase rated as 'success' | from the beginning to the end of colonoscopy (Baseline)
  Evaluate the overall cleanliness in four steps according to the results of each of the five colon sections Grade A: 3 or 4 points for all colon sections Grade B: One or more sections with a score of 2 Grade C: One or more sections with a score of 1 Grade D: One or more sections with a score of 0
  ※ If the overall colon cleanliness evaluation result is A grade, it is evaluated as successful 'failure (sealing success)' and C grade or D 'failure (sealing failure).

SECONDARY OUTCOMES:
Percentage of test subjects whose HCS cleanliness was evaluated as 'success' | from the beginning to the end of colonoscopy(Baseline)
  Evaluate the overall cleanliness in four steps according to the results of each of the five colon sections.
  Grade A: 3 or 4 points for all colon sections Grade B: One or more sections with a score of 2 Grade C: One or more sections with a score of 1 Grade D: One or more sections with a score of 0
  ※ If the overall colon cleanliness evaluation result is A grade, it is evaluated as successful 'failure (sealing success)' and C grade or D 'failure (sealing failure).
Overall cleanliness ratio on HCS (overall cleansing rate) | from the beginning to the end of colonoscopy(Baseline)
  Percentage of test subjects rated as grade A, B, C, and D on the HCS
Average score for each 5 compartments on the HCS (mean HCS score) | from the beginning to the end of colonoscopy(Baseline)
  Assessment of crystallinity by five colon sections (rector, sigmoid colon, descending colon, lateral colon, ascending colon)
Percentage of test subjects with residual air bubbles on the bubble score | from the beginning to the end of colonoscopy(Baseline)
  Assess the degree of gas removal (bubble degree) by five colon sections (rector, sigmoid colon, descending colon, lateral colon, ascending colon)
  Grade 0 No or minimal scattered bubbbles Grade 1 Bubbles covering at least half the luminal diameter Grade 2 Bubbles covering the circumference of the lumen Grade 3 Bubbles filling the entire lumen
Percentage of test subjects found to have polyps or adenoma (detection of polyp or adenoma) | from the beginning to the end of colonoscopy(Baseline)
  The examiner checks whether polyps or adenomas are found through colonoscopy, and the test subjects with one or more polyps/adenomas are defined as "detection."
Percentage of test subjects whose endoscopy has reached the appendix (cecal intubation rate) | from the beginning to the end of colonoscopy(Baseline)
  The cecal intubation is defined as passing the tip of a colonoscopy to the proximal part of the ileocecal valve so that the entire cecal caput is visible, including the inner wall of the cecal valve between the ileocecal valve and the cecal entrance
Total colonoscopy time | from the beginning to the end of colonoscopy(Baseline)
  The total colonoscopy time is the sum of colonoscopy insertion time and recovery time
Percentage of test subjects in taste category | End of colonoscopy(Baseline)
  Subsequently, the intention to use the same colon cleaner during colonoscopy is evaluated as "yes" and "no."
Percentage of subjects tested by compliance with administration of clinical trial drugs | End of colonoscopy(Baseline)
  1. Percentage of test subjects administered 100%
  2. Percentage of test subjects administered 75% or more and less than 100%
  3. Percentage of test subjects administered less than 75%
IP medication satisfaction | from the beginning to the end of colonoscopy(Baseline)
  (1) Average score of difficulty when taken
IP medication satisfaction | from the beginning to the end of colonoscopy(Baseline)
  (2) Percentage of test subjects in category of difficulty in taking
IP medication satisfaction | from the beginning to the end of colonoscopy(Baseline)
  (3) an average score of taste

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No